CLINICAL TRIAL: NCT01251926
Title: Pilot Study of Weekly EZN-2208 (Pegylated SN-38) in Combination With Bevacizumab in Refractory Solid Tumors
Brief Title: EZN-2208 (Pegylated SN-38) in Combination With Bevacizumab in Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110042; 11-C-0042; NCT01301547 (obsolete NCT alias)
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2014-05-02

CONDITIONS: Neoplasms
Keywords: Bevacizumab; Camptothecin; EZN-2208; Anti-Angiogenesis; Advanced Cancer; Cancer; Solid Tumor
MeSH Terms: conditions — Neoplasms | interventions — EZN-2208; Bevacizumab

INTERVENTIONS:
Drug: EZN-2208
Drug: Bevacizumab

SUMMARY:
Background:

- The anticancer drug bevacizumab works by reducing the formation of new blood vessels in tumors, which can slow or stop the growth of cancer cells and supporting blood vessels. The experimental drug EZN-2208 works by limiting how well cancer cells can divide. Drugs similar to EZN-2208 also work by turning off the production of the HIF protein, which otherwise can help cancer cells to grow even when blood supply is limited. Researchers are interested in determining if EZN-2208 turns off HIF in patient tumors, and whether combining it with bevacizumab is an effective treatment for cancers that have not responded to standard treatment.

Objectives:

- To assess the safety and effectiveness of the combination of EZN-2208 and bevacizumab for solid tumors that have not responded to standard treatment.

Eligibility:

- Individuals at least 18 years of age who have solid tumors that have not responded to standard treatment.

Design:

* Participants will be screened with a full physical examination and medical history, blood and urine samples, and tumor imaging studies.
* Participants will receive EZN-2208 and bevacizumab intravenously on an outpatient basis in 4-week cycles (with the exception of the first cycle, which will be 5 weeks).
* Cycle 1: Participants will receive EZN-2208 once a week for 3 weeks in a row (days 1, 8, and 15), followed by 1 week without the drug. Participants will receive bevacizumab 1 week before EZN-2208 (day - 7) and then 3 weeks later (day 15).
* Subsequent cycles: Participants will receive EZN-2208 once a week for 3 weeks in a row (days 1, 8, and 15), followed by 1 week without the drug. Participants will receive bevacizumab every 2 weeks (days 1 and 15).
* Participants will have clinic visits with physical examinations and blood tests in the first 3 weeks of each cycle. Clinic visits may also include tumor imaging studies and tumor biopsies as directed by the study researchers.
* Participants will continue to take the study drugs for as long as the tumor shrinks or does not grow, and as long as they do not experience intolerable or unsafe side effects from the drugs.

DETAILED DESCRIPTION:
Background

One reason postulated for the limited efficacy of anti-angiogenic or anti-VEGF agents such as bevacizumab is that they cause intra-tumoral hypoxia, resulting in the induction and up-regulation of hypoxia-inducible factors (HIF) such as HIF-1Alpha. These in turn play a central role in tumor progression by acting as master regulators of how cancer cells adapt to hypoxic conditions. HIF-1Alpha therefore represents an attractive target in oncology.

Camptothecin analogues (including SN-38, topotecan, and irinotecan) have been shown to consistently reduce the translation, expression, and transcriptional activity of HIF-1Alpha in vitro and in vivo, and therefore have the potential to inhibit the HIF-1? induction that occurs with anti-angiogenic agents.

The central rationale of this study is that HIF-1alpha induction by bevacizumab will be offset by weekly administration of EZN-2208 (PEGylated SN-38), and that this will result in synergistic anti-tumor effects.

Objectives

Determine the modulation of HIF-1alpha protein (by ELISA) in solid tumors after treatment with EZN-2208 and bevacizumab.

Determine the safety and tolerability of the combination of EZN-2208 and bevacizumab with EZN-2208 administered weekly times 3 (Days 1, 8, and 15) and bevacizumab administered every 2 weeks in 28-day cycles.

Perform correlative studies to assess changes in angiogenesis in tumor tissue.

Evaluate antitumor responses as determined by RECIST.

Eligibility

Adults with histologically documented solid tumors, whose disease has progressed following standard therapy or who have no acceptable standard treatment.

Performance status ECOG 0-2; adequate organ function; life expectancy at least 3 months; no major surgery, radiation or chemotherapy within 4 weeks prior to study enrollment; recovered from toxicities of prior therapies to at least eligibility levels.

Willingness to undergo tumor biopsies for research purposes.

Study Design

This is a single-arm pilot study.

Patients will receive EZN-2208 IV on Day 1, 8, and 15 of a 28-day cycle at a dose of 9 mg/m(2); bevacizumab will be administered IV every 2 weeks at a dose of 5 mg/kg.

For cycle 1: Bevacizumab will be administered on Day -7 (i.e., 1 week prior to EZN-2208) and Day 15.

For subsequent cycles: Bevacizumab will be administered on Day 1 and 15.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have histologically confirmed (by the Laboratory of Pathology, NCI) solid tumors that are metastatic or unresectable and for which standard therapies do not exist or are no longer effective.

There are no restrictions on prior therapy.

Age greater than or equal to18 years. Because no dosing or adverse event data are currently available on the use of EZN-2208 in combination with bevacizumab in patients less than 18 years of age, children are excluded from this study, but will be eligible for future pediatric Phase I combination trials.

ECOG performance status less than or equal to 2 (Karnofsky greater than or equal to 60%

Life expectancy of greater than 3 months.

Patients must have normal organ and marrow function as defined below:

leukocytes greater than or equal to 3,000/mcL

absolute neutrophil count greater than or equal to 1,500/mcL

platelets greater than or equal to 100,000/mcL

total bilirubin less than or equal to 1.5 times the institutional upper limit of normal

AST(SGOT)/ALT(SGPT) less than or equal to 2.5 times the institutional upper limit of normal

creatinine less than or equal to 1.5 times the institutional upper limit of normal

OR

creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.

The effects of EZN-2208 on the developing human fetus are unknown. For this reason and because bevacizumab is known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 3 months after completion of study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Ability to understand and the willingness to sign a written informed consent document.

Disease amenable to biopsy, and willingness to undergo biopsies.

EXCLUSION CRITERIA:

Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Patients must be (Bullet) 2 weeks since receiving study drug as a participant in a Phase 0 study (also referred to as an early Phase I study where a subtherapeutic dose of drug is administered).

Patients may not be receiving any other investigational agents.

Patients with a diagnosis of colorectal cancer, who have previously failed treatment with a topoisomerase I inhibitor. Patients with all other types of malignancies will be considered for eligibility regardless of prior exposure to topoisomerase 1 inhibitors.

History of allergic reactions attributed to compounds of similar chemical or biologic composition to EZN-2208 or bevacizumab.

Uncontrolled intercurrent illness including, but not limited to, clinically significant cardiovascular disease as defined below, or psychiatric illness/social situations that would limit compliance with study requirements.

Pregnant women are excluded from this study because bevacizumab is an antiangiogenic agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with EZN-2208, breastfeeding should be discontinued if the mother is treated with EZN-2208.

HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with EZN-2208. In addition, these patients are at increased risk of lethal infections when treated with marrowsuppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Urine protein should be screened by urine analysis. If protein is 2+ or higher, 24-hour urine protein should be obtained and the level should be <1000 mg for patient enrollment.

Serious or non-healing wound, ulcer, or bone fracture. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months.

Invasive procedures defined as follows:

* Major surgical procedure, open biopsy, or significant traumatic injury within the past 28 days.
* Anticipation of need for major surgical procedures during the course of the study.

Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within the past 6 months.

Known CNS disease except for treated brain metastasis. Treated brain metastases are defined as having no ongoing requirement for steroids and no evidence of progression or hemorrhage after treatment for at least 3 months, as ascertained by clinical examination and brain imaging (MRI or CT). Patients receiving EIAED anticonvulsants will not be eligible to participate (Appendix B). Patients on non-EIAED may be enrolled at the discretion of the PI. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent), or a combination as deemed appropriate by the treating physician.

Patients with clinically significant cardiovascular disease are excluded:

* Inadequately controlled hypertension (systolic blood pressure >160 mm Hg and/or diastolic blood pressure >90 mm Hg despite antihypertensive medication)
* History of stroke/cerebrovascular accident within 6 months
* Myocardial infarction or unstable angina within 6 months
* New York Heart Association grade II or greater congestive heart failure
* Serious and inadequately controlled cardiac arrhythmia
* Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection)
* Clinically significant peripheral vascular disease

Evidence of bleeding diathesis or coagulopathy. Patients on therapeutic anticoagulation will be excluded.

Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-11-15; Study Completion 2014-04-23 (Actual)

PRIMARY OUTCOMES:
Determine the modulation of HIF-1Alpha protein (by ELISA) in solid tumors after treatment with EZN-2208 and bevacizumab.

SECONDARY OUTCOMES:
Determine the safety and tolerability of the combination of EZN-2208 and bevacizumab with EZN-2208 administered weekly times 3 (Days 1, 8, and 15) and bevacizumab administered every 2 weeks in 28-day cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Semenza GL. Hypoxia and cancer. Cancer Metastasis Rev. 2007 Jun;26(2):223-4. doi: 10.1007/s10555-007-9058-y. No abstract available. PMID 17404692
- [Background] Jiang BH, Liu LZ. AKT signaling in regulating angiogenesis. Curr Cancer Drug Targets. 2008 Feb;8(1):19-26. doi: 10.2174/156800908783497122. PMID 18288940
- [Background] Presta LG, Chen H, O'Connor SJ, Chisholm V, Meng YG, Krummen L, Winkler M, Ferrara N. Humanization of an anti-vascular endothelial growth factor monoclonal antibody for the therapy of solid tumors and other disorders. Cancer Res. 1997 Oct 15;57(20):4593-9. PMID 9377574